CLINICAL TRIAL: NCT06575933
Title: A Study to Evaluate the Effect of Single and Multiple Doses of MK-1084 on the Single-Dose Pharmacokinetics of Midazolam and Digoxin in Healthy Participants
Brief Title: A Study of Calderasib (MK-1084) With Midazolam and Digoxin in Healthy Participants (MK-1084-009)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 1084-009; CA43815 (Other: Celerion Protocol Number); MK-1084-009 (Other: MSD)
Record Dates: First submitted 2024-08-26; First posted 2024-08-28 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Non-small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Midazolam; Digoxin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Period 1: Midazolam and Digoxin (Experimental): Participants will receive a single oral dose of midazolam and a single oral dose of digoxin on Day 1.
  Interventions: Drug: Midazolam; Drug: Digoxin
- Period 2: Calderasib, Midazolam, and Digoxin (Experimental): A washout period of at least 10 days will occur following midazolam and digoxin dosing in Period 1 and the first calderasib dosing in Period 2. Participants will receive calderasib once daily on Days 1 through Day 15 with a single oral dose of midazolam on Days 1, 6, and 14 and a single oral dose of digoxin on Days 1 and 11.
  Interventions: Drug: Calderasib; Drug: Midazolam; Drug: Digoxin

INTERVENTIONS:
Drug: Calderasib — Oral administration
  Other Names: MK-1084
  Arms: Period 2: Calderasib, Midazolam, and Digoxin
Drug: Midazolam — Oral administration
Drug: Digoxin — Oral administration

SUMMARY:
The goal of the study is to see what happens to levels of midazolam and digoxin in a person's body over time (a pharmacokinetic or PK study). Researchers will compare what happens to midazolam and digoxin in the body when it is given with and without another medicine called calderasib. Researchers are testing if digoxin and midazolam levels in the body are different when digoxin and midazolam are given with or without calderasib.

ELIGIBILITY:
Inclusion Criteria:

The key inclusion criteria include but are not limited to the following:

* Is medically healthy with no clinically significant medical history, physical examination, laboratory profiles, vitals signs, and electrocardiograms (ECGs)
* Has a body mass index (BMI) ≥18 and ≤32 kg/m^2, inclusive

Exclusion Criteria:

The key exclusion criteria include but are not limited to the following:

* Has a medical history that may confound the results of the study or poses an additional risk to the participant in the study
* Has a history or presence of hypersensitivity or idiosyncratic reaction to the study drugs or related compounds

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2024-09-03 (Actual); Primary Completion 2024-10-28 (Actual); Study Completion 2024-10-28 (Actual)

PRIMARY OUTCOMES:
Area Under the Concentration-Time Curve from Time 0 to Infinity (AUC0-Inf) of Midazolam | Predose and at designated timepoints up to 24 hours postdose
  Blood samples will be collected to determine the AUC0-inf of midazolam.
Area Under the Concentration-Time Curve from Time 0 to Last (AUC0-Last) of Midazolam | Predose and at designated timepoints up to 24 hours postdose
  Blood samples will be collected to determine the AUC0-last of midazolam.
Area Under the Concentration-Time Curve from Time 0 to 24 hours (AUC0-24hr) of Midazolam | Predose and at designated timepoints up to 24 hours postdose
  Blood samples will be collected to determine the AUC0-24hr of midazolam.
Maximum Plasma Concentration (Cmax) of Midazolam | Predose and at designated timepoints up to 24 hours postdose
  Blood samples will be collected to determine the Cmax of midazolam.
Time to Maximum Plasma Concentration (Tmax) of Midazolam | Predose and at designated timepoints up to 24 hours postdose
  Blood samples will be collected to determine the Tmax of midazolam.
Apparent Terminal Half-life (t1/2) of Midazolam | Predose and at designated timepoints up to 24 hours postdose
  Blood samples will be collected to determine the t1/2 of midazolam.
Apparent Clearance (CL/F) of Midazolam | Predose and at designated timepoints up to 24 hours postdose
  Blood samples will be collected to determine the CL/F of midazolam.
Apparent Volume of Distribution During Terminal Phase (Vz/F) of Midazolam | Predose and at designated timepoints up to 24 hours postdose
  Blood samples will be collected to determine the Vz/F of midazolam.
AUC0-Inf of Digoxin | Predose and at designated timepoints up to 120 hours postdose
  Blood samples will be collected to determine the AUC0-inf of digoxin.
AUC0-Last of Digoxin | Predose and at designated timepoints up to 120 hours postdose
  Blood samples will be collected to determine the AUC0-last of digoxin.
AUC0-24hr of Digoxin | Predose and at designated timepoints up to 24 hours postdose
  Blood samples will be collected to determine the AUC0-24hr of digoxin.
Cmax of Digoxin | Predose and at designated timepoints up to 120 hours postdose
  Blood samples will be collected to determine the Cmax of digoxin.
Tmax of Digoxin | Predose and at designated timepoints up to 120 hours postdose
  Blood samples will be collected to determine the Tmax of digoxin.
t1/2 of Digoxin | Predose and at designated timepoints up to 120 hours postdose
  Blood samples will be collected to determine the t1/2 of digoxin.
CL/F of Digoxin | Predose and at designated timepoints up to 120 hours postdose
  Blood samples will be collected to determine the CL/F of digoxin.
Vz/F of Digoxin | Predose and at designated timepoints up to 120 hours postdose
  Blood samples will be collected to determine the Vz/F of digoxin.

SECONDARY OUTCOMES:
AUC0-24hr of Calderasib | Predose and at designated timepoints up to 24 hours postdose
  Blood samples will be collected to determine the AUC0-24hr of calderasib.
AUC0-Last of Calderasib | Predose and at designated timepoints up to 24 hours postdose
  Blood samples will be collected to determine the AUC0-last of calderasib.
Cmax of Calderasib | Predose and at designated timepoints up to 24 hours postdose
  Blood samples will be collected to determine the Cmax of calderasib.
C24 of Calderasib | Predose and at designated timepoints up to 24 hours postdose
  Blood samples will be collected to determine the Cmax of calderasib.
Tmax of Calderasib | Predose and at designated timepoints up to 24 hours postdose
  Blood samples will be collected to determine the Tmax of calderasib.
t1/2 of Calderasib | Predose and at designated timepoints up to 24 hours postdose
  Blood samples will be collected to determine the t1/2 of calderasib.
Cmax Accumulation Ratio of Calderasib | Predose and at designated timepoints up to 24 hours postdose
  Blood samples will be collected to determine the Cmax accumulation ratio of calderasib. The accumulation ratio is the ratio of Predose Cmax to the 24 hour Cmax
AUC0-24 Accumulation Ratio of Calderasib | Predose and at designated timepoints up to 24 hours postdose
  Blood samples will be collected to determine the AUC0-24 accumulation ratio of calderasib. The accumulation ratio is the ratio of Predose AUC0-24 to the 24 hour AUC0-24.
Amount of Drug Excreted in Urine from Time 1 to Time 2 (Aet1-t2) of Digoxin | Predose and at designated timepoints up to 120 hours postdose
  Urine samples will be collected to determine the Aet1-t2 of digoxin.
Total Amount of Drug Excreted in Urine (Ae) of Digoxin | Predose and at designated timepoints up to 120 hours postdose
  Urine samples will be collected to determine the Ae of digoxin.
Fraction of Unchanged Digoxin in Urine (Fe) | Predose and at designated timepoints up to 120 hours postdose
  Urine samples will be collected to determine the Fe of digoxin.
Number of Participants Who Experience an Adverse Event (AE) | Up to approximately 1 month
  An AE is any untoward medical occurrence in a participant, temporally associated with the use of study treatment, whether or not considered related to the study treatment. The number of participants who experience an AE will be reported.
Number of Participants Who Discontinue Study Due to an AE | Up to approximately 1 month
  An AE is any untoward medical occurrence in a participant, temporally associated with the use of study treatment, whether or not considered related to the study treatment. The number of participants who discontinue study due to an AE will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (1):
- Celerion ( Site 0001), Tempe, Arizona, United States

IPD SHARING:
Plan to Share IPD: Yes
https://trialstransparency.msdclinicaltrials.com/pdf/ProcedureAccessClinicalTrialData.pdf
URL: https://externaldatasharing-msd.com/

REFERENCES:
- See also: Merck Clinical Trials Information — https://www.merckclinicaltrials.com/